CLINICAL TRIAL: NCT02931591
Title: Effect of Insulin Sensitization on Insulin Like Growth Factor-1 Responses to Growth Hormone Treatment in Children Born Small for Gestational Age
Brief Title: Effect of Insulin Sensitization on IGF-1 Response to Growth Hormone in SGA Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Rigshospitalet, Denmark (Other); Birmingham Women's and Children's NHS Foundation Trust (Other); The National Children's Hospital, Tallaght (Other)
Responsible Party: Principal Investigator, David B Dunger, Professor of Paediatrics, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGA Metformin Study
Record Dates: First submitted 2016-09-14; First posted 2016-10-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Small for Gestational Age
Keywords: Small for gestational age; insulin sensitivity; IGF-1 response; growth hormone treatment
MeSH Terms: conditions — Insulin Resistance | interventions — Metformin; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GH+Metformin (Active Comparator): The children will be given both Growth Hormone and Metformin for 6 months
  Interventions: Drug: Metformin; Drug: Growth Hormone
- GH+Placebo (Placebo Comparator): Children will be given both GH and Placebo for 6 months
  Interventions: Drug: Growth Hormone; Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin is administered as an oral solution
  Arms: GH+Metformin
Drug: Growth Hormone — Growth Hormone- no specific band
Drug: Placebo
  Arms: GH+Placebo

SUMMARY:
This study is aimed to determine if Metformin treatment in children born small for gestational age (SGA) who are being treated with Growth Hormone (GH) for short stature improves the response to GH by producing greater concentrations of Insulin-like growth factor -1 (IGF-1) in the blood.

DETAILED DESCRIPTION:
Growth hormone treatment (GH) is recommended in children born small for gestational age (SGA) who fail to catch-up. SGA is a heterogeneous condition as reflected in the varied response to GH treatment. Variable generation and resistance to Insulin-like growth factor-1 (IGF-1), the most important circulating mediator of GH action may underpin this heterogeneity. An association between the variants in the genes related to lower insulin sensitivity and reduced IGF-1 and growth response to GH therapy in SGA children have been reported recently. The hypothesis of this study is that insulin sensitivity may be causally linked to the response to GH therapy, and adjuvant therapy with an insulin sensitizer may improve IGF-1 generation, decrease IGF-I resistance and optimise growth response.

To explore this hypothesis, this study aims to determine the effects of insulin sensitization using Metformin as an adjuvant to a fixed dose GH therapy for 6 months in short SGA children. The patients will be short SGA children between age 4 -10 years and identified from three paediatric endocrine units in Denmark, Ireland and the United Kingdom. In this mechanistic study 24 subjects starting GH treatment will be randomised in a 1:1 ratio to adjunctive Metformin or placebo for 6 months and followed-up for another 6months. The participants will receive GH treatment for the entire duration of the study (12 months) and will undergo an oral glucose tolerance test and dual-energy x-ray absorptiometry scan to determine glucose metabolism and body fat mass respectively at baseline and 6 months, and will have 3 monthly measurements of height, weight and skinfold thickness. The primary outcome will be the area under the curve of IGF-1 levels measured at 0, 1, 3 and 6 months. Secondary outcomes will include changes in insulin sensitivity, height, body fat mass and safety measures at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* SGA children eligible for GH treatment according to European Medicines Agency (EMA) and The National Institute for Health and Care Excellence (NICE) criteria
* Gestational age at birth >28 weeks
* Age 4-9 years in girls and 4-10 years in boys
* Prepubertal at start of treatment
* Naïve to GH therapy

Exclusion Criteria:

* Known or suspected allergy to GH
* Previous participation in a GH trial
* Severe learning difficulties
* Previous or active malignancy
* Benign intracranial hypertension

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
IGF-1 response | 6 months
  Area under the curve of IGF-1 standard deviation scores over 6 months

SECONDARY OUTCOMES:
Height velocity | 6 months and 1 year
  Height increments
Insulin sensitivity | 6 months and 1 year
  Measured by homeostasis model assessment model
Insulin secretion | 6 months
  Measured by oral glucose tolerance test

IPD SHARING:
Plan to Share IPD: No